CLINICAL TRIAL: NCT04573491
Title: Implementation of Pharmacogenetic Testing as Part of Medication Reviews in Hospital Wards
Brief Title: Implementation of Pharmacogenetic Testing in Hospital Wards
Acronym: FAGLIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pharmacy Enterprise, South Eastern Norway (Other)
Collaborators: University Hospital, Akershus (Other); Diakonhjemmet Hospital (Other); University of Oslo School of Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMP-CYP SA HF 2020-001
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Admitted Multimorbid Patients
Keywords: pharmacogenetics; implementation; medication review
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacogenetic test (Experimental): Medication review including results from pharmacogenetic testing
  Interventions: Genetic: Pharmacogenetic test; Other: Medication review

INTERVENTIONS:
Genetic: Pharmacogenetic test — genotyping for genes that affect drug metabolism
Other: Medication review — systematic and interdisciplinary method aiming to increase quality of medication treatment

SUMMARY:
The purpose of this study is to investigate whether it is feasible to implement pharmacogenetic testing as part of medication review while the patient is admitted to hospital.

DETAILED DESCRIPTION:
Earlier studies have shown that pharmacogenetic testing may contribute to optimizing the efficacy of medication treatment and to reduce the risk of adverse effects. Inclusion of pharmacogenetic testing as part of medication reviews reveals more serious drug related problems and leads to more changes in medication treatment than medication review alone.

The use of pharmacogenetic testing as part of medication reviews has not earlier been systematically investigated in hospital patients in Norway. There is little documentation of what is needed to implement the use of pharmacogenetic testing in a hospital ward.

The investigators are conducting a descriptive study in two internal medicine wards at Akershus University Hospital. 50 patients using minimum 5 regular drugs including at least one relevant for pharmacogenetic testing will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 long-term conditions
* at least 5 regular drugs of which at least one relevant for pharmacogenetic testing
* at least 2 years life expectancy
* able to communicate in Norwegian
* able to give informed consent
* summary care record

Exclusion Criteria:

* moderate to severe dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with results from pharmacogenetic testing included in medication review | from admission to discharge, an average of 1 week
  Number of patients

SECONDARY OUTCOMES:
Acceptance of recommendations | after medication review and before discharge, an average of 3 days
  Degree of acceptance of recommendations after pharmacogenetic testing, by prescribers
Documentation of information from pharmacogenetic testing | after medication review and before discharge, an average of 3 days
  Number of patients with information from pharmacogenetic testing documented in the patient journal

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Bjerknes, Ph.D, Study Director — Hospital Pharmacy Enterprise, South Eastern Norway
Locations (1):
- Akershus University Hospital, Lørenskog, Nordbyhagen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hjemas BJ, Bovre K, Bjerknes K, Mathiesen L, Mellingsaeter MCR, Molden E. Implementation of pharmacogenetic testing in medication reviews in a hospital setting. Br J Clin Pharmacol. 2023 Oct;89(10):3116-3125. doi: 10.1111/bcp.15815. Epub 2023 Jun 22. PMID 37277227